CLINICAL TRIAL: NCT04691908
Title: Multicenter, Randomized, Blind, Placebo-controlled Clinical Study of III Phase on Assessment of Preventive Efficiency, Safety and Immunogenicity QazCovid-in®-Vaccine Against COVID-19 in Healthy Adult Volunteers
Brief Title: Immunogenicity, Efficacy and Safety of QazCovid-in® COVID-19 Vaccine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Research Institute for Biological Safety Problems (Other Government)
Collaborators: City polyclinic No. 4 of the of Almaty Ministry of Healthcare of the Republic of Kazakhstan (Unknown); Clinic of the International Institute of Postgraduate Education Ministry of Healthcare of the Republic of Kazakhstan (Unknown); City Multidisciplinary Hospital of Zhambyl Region Ministry of Healthcare of the Republic of Kazakhstan (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: QAZCOV-III-01/2020
Record Dates: First submitted 2020-12-21; First posted 2020-12-31 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Covid19; SARS-CoV Infection; Vaccine Adverse Reaction
Keywords: QazCovid-in®, vaccine, III phase, efficiency, safety, immunogenicity
MeSH Terms: conditions — COVID-19; Severe Acute Respiratory Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phase III Adult-vaccine (A Sample, blind study) (Active Comparator): Group 1 (phase III): 2400 volunteers from 18 years old and elder who will be the QazCovid-in® twice spaced 21 days apart, intramuscularly, at a dose of 0.5 ml
  Interventions: Biological: QazCovid-in®-vaccine against COVID-19
- Phase III Adult-Placebo (A Sample, blind study) (Placebo Comparator): Group 1 (phase III): 600 volunteers from 18 years old and elder who will be the Placebo twice spaced 21 days apart, intramuscularly, at a dose of 0.5 ml
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: QazCovid-in®-vaccine against COVID-19 — QazCovid-in® (inactivated) Vaccine manufactured by Research Institute for Biological Safety Problems Republic of Kazakhstan
  Arms: Phase III Adult-vaccine (A Sample, blind study)
Other: Placebo — Placebo (sodium chloride buffs, solvent for the preparation of dosage forms for injection 0.9%)
  Arms: Phase III Adult-Placebo (A Sample, blind study)

SUMMARY:
Multicenter, randomized, blind, placebo-controlled clinical study of III phases on the assessment of preventive efficiency, safety and immunogenicity QazCovid-in®-vaccine against COVID-19 in healthy adult volunteers

DETAILED DESCRIPTION:
The main objective of the study is to prove the superiority of the QazCovid-in®-vaccine inactivated against COVID-19 in comparison with placebo in terms of seroconversion (the proportion of persons with a fourfold or higher increase in antibody titers to SARS-CoV-2) on the 21st, 42nd day, 90th and 180th days after vaccination.

To evaluate the immunogenicity of the QazCovid-in® vaccine inactivated against COVID-19 versus placebo.

Evaluate vaccine efficacy.

Evaluate the safety of vaccine versus placebo.

ELIGIBILITY:
Inclusion Criteria:

Availability of signed and dated informed consent of the volunteer to participate in the study.

Healthy male and female volunteers aged 18 and above. Ability and voluntary desire to independently keep records in the Self-Observation Diary, as well as to carry out all the repeated visits provided for in the study for control medical observation.

The voluntary desire of females to use methods of reliable contraception throughout the entire period of their participation in the study.

Negative results for IgM and IgG antibodies to SARS-CoV-2. Absence of COVID-19 diagnosis in history. Absence in the last 14 days of close contact with persons suspected of being infected with SARS-CoV-2, or persons whose diagnosis of COVID-19 has been confirmed with laboratory.

Exclusion Criteria:

Aggravated allergic history, drug intolerance, including hypersensitivity to any of the components of the study drug, as well as a history of serious adverse events during vaccine administration (such as allergic reactions, respiratory failure, angioedema, abdominal pain).

Acute illness with a fever (body temperature ≥37.1 ° C) at the time of screening.

History of chronic alcohol abuse and/or drug use. Positive results for antibodies IgM, IgG to SARS-CoV-2 Women with a positive urine pregnancy test. Simultaneous treatment with immunosuppressive drugs, incl. corticosteroids (2 weeks) 4 weeks prior to study drug administration.

Acute or chronic clinically significant lesions of the lungs, cardiovascular system, gastrointestinal tract, liver, blood system, skin, endocrine, neurological and psychiatric diseases or impaired renal function (asthma, diabetes, thyroid disease, arrhythmia, heart attack myocardium, severe hypertension not controlled by drugs, etc.), identified based on the data of the medical history, physical examination, which, according to the researcher, may affect the study result.

History of platelet disorder or other blood clotting disorders that may cause contraindications to intramuscular administration.

History of leukemia or neoplasm. Persons with autoimmune diseases. A history of Guillain-Barré syndrome or other neuroimmunological diseases. Subjects who received antiviral drugs, immunoglobulins or blood transfusions or any other investigational drug within 4 weeks prior to study drug administration; Subjects who received anti-inflammatory drugs 2 days prior to study drug administration; Participation in any other clinical research within the last 6 months. Subjects with regard to whom there is a concern that they will not comply with the requirements of the study, or persons with severe physical or mental disabilities that may affect the completion of the study.

Voluntary refusal to study. Vulnerable research subjects.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3000 (Actual)
Dates: Start 2020-12-25 (Actual); Primary Completion 2021-04-26 (Actual); Study Completion 2021-07-11 (Actual)

PRIMARY OUTCOMES:
Terms of seroconversion (the proportion of persons with a fourfold or higher change in antibody titers to SARS-CoV-2) | at days 0, 21, 42, 90, 180
  The main objective of the study is to prove the superiority of the QazCovid-in®-vaccine inactivated against COVID-19 in comparison with placebo in terms of seroconversion (the proportion of persons with a fourfold or higher change in antibody titers to SARS-CoV-2)
To evaluate the immunogenicity of the QazCovid-in® vaccine inactivated against COVID-19 versus placebo | at days 0, 21, 42, 90, 180
  The geometric mean titer of serum antibodies ELISA to SARS-CoV-2 after vaccination. The multiplicity of the change in the geometric mean titer of serum antibodies to SARS-CoV-2 after vaccination.
Frequency of confirmed cases of COVID-19 | through study completion, an average of 6 months
  The presence of clinical manifestations and a positive laboratory test for SARS-CoV-2 virus RNA within 6 months after vaccination

SECONDARY OUTCOMES:
Changing of antigen-specific cellular immunity level | at days 0, 90, 180
  Determination of the level of production of intracellular cytokines by antigen-activated T-lymphocytes
Frequency of adverse events up to seven days after immunization | Seven days after each immunization
  Frequency of adverse reaction in the seven days following each immunization per age group
Frequency of adverse events up to 21 days after immunization | 21 days after each immunization
  Frequency of adverse reaction in the 21 days following each immunization per age group
Incidence of serious adverse events during the study | throughout the study, an average of 6 months
  Incidence of serious adverse events during the study

CONTACTS AND LOCATIONS:
Overall Officials: Berik Khairullin, PhD, Study Director — Research Institute for Biological Safety Problems Committee of Science of the Ministry of Education and Science of the Republic of Kazakhstan; Kunsulu Zakarya, PhD, Study Chair — Research Institute for Biological Safety Problems Committee of Science of the Ministry of Education and Science of the Republic of Kazakhstan; IIlyas Kulmagambetov, PhD, Principal Investigator — Centre for Clinical Medicine and Research
Locations (1):
- Research Institute for Biological Safety Problems Committee of Science of the Ministry of Education and Science of the Republic of Kazakhstan, Gvardeyskiy, Jambul, Kazakhstan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Khairullin B, Zakarya K, Orynbayev M, Abduraimov Y, Kassenov M, Sarsenbayeva G, Sultankulova K, Chervyakova O, Myrzakhmetova B, Nakhanov A, Nurpeisova A, Zhugunissov K, Assanzhanova N, Nurabayev S, Kerimbayev A, Yershebulov Z, Burashev Y, Kulmagambetov I, Davlyatshin T, Sergeeva M, Buzitskaya Z, Stukova M, Kutumbetov L. Efficacy and safety of an inactivated whole-virion vaccine against COVID-19, QazCovid-in(R), in healthy adults: A multicentre, randomised, single-blind, placebo-controlled phase 3 clinical trial with a 6-month follow-up. EClinicalMedicine. 2022 Jun 25;50:101526. doi: 10.1016/j.eclinm.2022.101526. eCollection 2022 Aug. PMID 35770251